CLINICAL TRIAL: NCT05163431
Title: Dimensional Validation of the Hallux Valgus Orthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Orthèse Hallux Valgus Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-19-0241_HV_HV
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Painful Hallux Valgus (Experimental)
  Interventions: Device: Hallux Valgus orthosis

INTERVENTIONS:
Device: Hallux Valgus orthosis — Custom designed orthosis and manufactured by 3D printing.

SUMMARY:
The goal of this project is to optimize the design of the orthosis by establishing the key volumetric characteristics of the custom iterations in order to subsequently transpose them to a standard model and establish the increment proportions of the different sizes. The final product should reduce the pain by repositioning the phalanges of the first toe with the first metatarsal in its axis.

ELIGIBILITY:
Inclusion Criteria:

* Painful hallux valgus
* three people maximum per shoe size

Exclusion Criteria:

* People with diabetes ;
* People with severe obesity ;
* People with hallux rigidus;
* People wearing full-time foot orthosis;
* People wearing high heel shoes regularly ;
* People with degenerative disease ;
* People with neuromuscular pathology ;
* People with a circulatory disorder ;
* People who have had major lower body surgery;
* People with epilepsy or with a history of epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in big toe deviation angle during gait at 1 month | At baseline and 1 month
  The big toe deviation angle is the angle between the big toe and the gait axis and measured with a motion capture system.
Change in pain at 1 month | At baseline and 1 month
  Pain is measured with a Likert scale from 1 (decrease of pain) to 5 (increase of pain).
Change in comfort at 1 month | At baseline and 1 month
  Comfort is measured with a Likert scale from 1 (not comfortable) to 5 (very comfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Edith Martin, PhD, Principal Investigator — TOPMED
Locations (1):
- TOPMED, Québec, Quebec, Canada